CLINICAL TRIAL: NCT06879834
Title: Assessing of Artificial Intelligence-based Software Platform for Diabetic Retinopathy Screening
Acronym: ARTDR
Status: Recruiting | Type: Observational
Sponsor: The Filatov Institute of Eye Diseases and Tissue Therapy (Other)
Collaborators: CheckEye LLC (Industry); Oftacentro SA (Other)
Responsible Party: Principal Investigator, Andrii Korol, MD, PhD, MD, PhD, DMedSc,Prof, The Filatov Institute of Eye Diseases and Tissue Therapy
Other Study IDs: 02.10.2024
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic Retinopathy; Fundus photo; nonmydriatic camera; Artificail Intelligence; CheckEye; Fundus image; fundus photography
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- main group: have diabetes mellitus
  Interventions: Device: taking fundus photos using non-mydriatic fundus camera
- control group: have risk factors for developing diabetes mellitus
  Interventions: Device: taking fundus photos using non-mydriatic fundus camera

INTERVENTIONS:
Device: taking fundus photos using non-mydriatic fundus camera — using artificial intelligence to identify diabetic retinopathy in the early stages using fundus photography.

SUMMARY:
To examine the potential for the detection of diabetic retinopathy (DR) using the artificial intelligence (AI)-based software platform Retina-AI.

DETAILED DESCRIPTION:
Operator took fundus images with a non-mydriatic fundus camera as per the Retina-AI CheckEye imaging protocol (an optic disc centered image and a fovea centered image for each eye).Thereafter, operator uploaded fundus images in the AI system for processing by the neural network.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of diabetes mellitus by definition.
2. Understanding of the Study and willingness and ability to sign informed consent
3. Patient age 18 or above
4. Diagnostic for diabetes: 4a) Type 1 diabetes of a lest 5 years of evolution; or 4b) Type 2 diabetes

Exclusion Criteria:

-1. Patients under 18 years of age; 2. Failure to give informed consent; 3. Presence of retinal diseases - acquired disease: age-related macular degeneration (AMD), occlusion of retinal vessels (ORV), etc.; birth defects: coloboma of choroid or optic nerve disc, etc.; hereditary diseases: retinitis pigmentosa, angioid streaks of the retina, etc.

4. A patient who has already undergone treatment (surgery, laser, etc.) for any disease of the retina: age-related macular degeneration (AMD), retinal vascular occlusion (ARV), etc. These patients should be excluded or allocated to a separate group.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 participants were planed to include in study, 100 of them had diabetes mellitus and 100 participants were as a control group have risk factors for diabetes mellitus.
  All participants were selected for the study based on the following inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-02 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The accuracy | Baseline
  The accuracy of detecting of DR

SECONDARY OUTCOMES:
The percent of invalid images | Baseline
  The percent of invalid images for analysing by neural network
The percent of false positive detection of DR | Baseline
  The percent of false positive detection of DR in individuals without DR

CONTACTS AND LOCATIONS:
Overall Officials: Andrii MD Korol, PhD, Principal Investigator — The Filatov Institute of Eye Diseases and Tissue Therapy
Locations (1):
- The Filatov Institute of Eye Diseases and Tissue Therapy, Odesa, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Detecting diabetic retinopathy using an artificial intelligence-based software platform: a pilot study — https://ua.ozhurnal.com/index.php/files/article/view/101